CLINICAL TRIAL: NCT03265054
Title: Evaluation of the Predictive Value of the Microvesicle Coagulo-lytic Balance in the Recurrence of Venous Thrombosis
Acronym: MICROREVE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-04
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Venous Thromboembolism (VTE)
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- re-thrombosis: adult patients with a VTE history with at least 3 months of anticoagulant treatment, which suffered from a re-thrombosis within 5 years after stopping the anticoagulant treatment
  Interventions: Biological: Analysis of plasma samples
- no thrombosis recurrence: adult patients with a VTE history with at least 3 months of anticoagulant treatment, without thrombosis recurrence
  Interventions: Biological: Analysis of plasma samples

INTERVENTIONS:
Biological: Analysis of plasma samples — Measuring microparticles (MPs) in Human Plasma Samples

SUMMARY:
Venous thromboembolism (VTE) including deep vein thrombosis (DVT) and pulmonary embolism (PE) affects about 1,200,000 individuals each year in Europe. About 50% of VTE are unprovoked and 20% of these patients will face a recurrent event after the usual three to six-month course of anticoagulant treatment. To date, most patients are given prolonged anticoagulant treatment. However, anticoagulant treatment are associated with a major risk of bleeding (3%/year). Thus an accurate identification of patients with unprovoked VTE with a low risk of recurrence is needed to avoid unnecessary anticoagulant treatment with a risk of bleeding.

Over the past few years, microparticles (MPs) which are small vesicles originating from the budding of cellular membranes have emerged as important biological entities regulating hemostasis. MPs expose at their surface procoagulant molecules such as phosphatidylserin and tissue factor (TF). All data obtained in mouse models support a role of MPs in venous thrombosis mediated by the TF activation. Moreover, results from clinical studies showed that TF-MPs was associated with the risk of venous thrombosis. However, the predictive value of TF-MPs in the recurrence of VTE is unknown. Besides, no study has taken into account the recent progresses in the understanding of the role of MPs in haemostasis. Indeed, MPs vectorize molecules which are not only procoagulant but also profibrinolytic. The net result depends on a balance between both activities (the coagulo-lytic balance). This balance is can be measured by two complimentary assays on MPs.

We hypothesized that the coagu-lytic balance of MPs is associated with an increased risk of VTE recurrence after stopping the anticoagulant treatment.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with a VTE history with at least 3 months of anticoagulant treatment.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 adult patients with a VTE history with at least 3 months of anticoagulant treatment. 150 patients which suffered from a re-thrombosis within 5 years after stopping the anticoagulant treatment, will be age- and sex-matched with 150 without thrombosis recurrence.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
coagu-lytic balance of MPs | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France